CLINICAL TRIAL: NCT07014319
Title: Maribavir Treatment of Cytomegalovirus for Lymphoid Malignancy Patients Undergoing Bispecific Antibodies
Brief Title: Phase II Trial of Maribavir for CMV in Patients With Lymphoid Malignancy on Bispecific Antibodies
Acronym: MALMBA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, JaMin Byun, Professor, MD, PhD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2505-076-1641
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-06

CONDITIONS: Cytomegalovirus (CMV)
Keywords: CMV; MM; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — maribavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maribavir arm (Experimental): The Maribavir arm includes patients with a confirmed diagnosis of multiple myeloma, follicular lymphoma, or large B-cell lymphomas (including diffuse large B-cell lymphoma, high-grade B-cell lymphoma, transformed follicular lymphoma, or transformed marginal zone lymphoma) who are receiving bispecific antibody therapy. Patients must have documented clinically significant CMV infection, defined by either CMV end-organ disease or initiation of pre-emptive therapy based on plasma CMV viremia ≥ 500 IU/mL in two consecutive assessments and relevant clinical findings.
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Participants will receive maribavir 400 mg twice daily starting from Week 1 and continuing until clearance of CMV. CMV clearance is defined as either an unquantifiable plasma CMV DNA titer (i.e., below the lower limit of quantification [LLOQ]) as assessed by the local laboratory, or a CMV DNA level below 500 IU/mL in plasma without evidence of CMV disease.

SUMMARY:
This is an open-label, single arm, multicenter study to evaluate the feasibility of maribavir treatment in multiple myeloma and lymphoma patients undergoing bispecific antibody treatment and experiencing treatment emergent CMV events

DETAILED DESCRIPTION:
This open-label, single-arm, multicenter study aims to evaluate the safety and feasibility of maribavir in patients with multiple myeloma or lymphoma who develop cytomegalovirus (CMV) reactivation during bispecific antibody (BsAb) therapy. While BsAbs are increasingly used in lymphoma and multiple myeloma due to their high efficacy, they are associated with a high risk of infections, particularly CMV, especially in heavily pretreated and immunocompromised patients. Existing anti-CMV treatments are often limited by toxicity and accessibility. Maribavir, an oral antiviral with a novel mechanism and favorable safety profile, offers a promising alternative. Given the high CMV burden observed in this population, this study seeks to address an important unmet need.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥19 years of age at the time of signing the informed consent form (ICF).

  * Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures.

    ③ Subject is willing and able to adhere to the study visit schedule and protocol requirements.

    ④ Subject has documented diagnosis of multiple myeloma, follicular lymphoma, or large B-cell lymphoma (including diffuse large B-cell lymphoma, high-grade B-cell lymphoma, transformed follicular lymphoma, or transformed marginal zone lymphoma), and is receiving one of the following bispecific antibodies: Multiple Myeloma: Teclistamab, Elranatamab, Talquetamab, Cevostamab, ABBV383 Lymphomas: Mosunetuzumab, Glofitamab, Epcoritamab, Odronextamab

    ⑤ Subject has documented clinically significant CMV infection, defined as: A. Onset of CMV end-organ disease (Appendix 1), or B. Initiation of anti-CMV pre-emptive therapy based on documented CMV viremia ≥500 IU/mL in two consecutive assessments (≥1 day apart) and the clinical condition of the subject Note: Prior therapy with ganciclovir, valganciclovir, foscarnet, or cidofovir is allowed.
    * ECOG performance status of 0, 1, or 2. ⑦ Individual of childbearing potential (IOCBP) must: A. Have two negative pregnancy tests before study treatment, and agree to ongoing testing.

B. Commit to true abstinence or use two forms of contraception (one highly effective + one barrier method) starting 28 days prior to treatment, during treatment, and for 90 days after the last dose.

Note: Definition of IOCBP includes menstruating individuals who are not postmenopausal for 12+ months or have not undergone permanent sterilization.

⑧ Male subjects must: A. Practice true abstinence (monthly verified) or use a condom with partners who are pregnant or of childbearing potential during treatment, dose interruptions, and for 90 days after last dose, regardless of vasectomy status.

⑨ Male subjects must not donate sperm during treatment and for 90 days after the last dose.

⑩ Female subjects must not donate eggs during treatment and for 90 days after the last dose.

Exclusion Criteria:

* Requires ganciclovir, valganciclovir, foscarnet, or cidofovir for non-CMV indications or requires co-administration with maribavir.

  * Known hypersensitivity to maribavir. ③ CMV disease involving the CNS (retinitis alone is allowed). ④ Received allogeneic SCT within 1 year or autologous SCT within 12 weeks prior to study treatment.

Allogeneic SCT recipients must not have active GVHD. ⑤ Any significant medical condition, infection, lab abnormality, or psychiatric illness posing unacceptable risk.

* Any condition that may confound data interpretation. ⑦ Any of the following laboratory abnormalities:

A. Creatinine clearance <10 mL/min or requiring dialysis (Cockcroft-Gault formula used):

* Males: CrCl = (140 - age) × weight (kg) / (72 × creatinine [mg/dL])
* Females: Multiply above result by 0.85 B. AST or ALT >5 × ULN C. Total bilirubin >3 × ULN (except Gilbert's syndrome)

  * Gastrointestinal disease or surgery (e.g., gastric bypass) that affects maribavir absorption.

    * Severe vomiting, diarrhea, or GI illness within 24 hours before first dose. ⑩ Use of immunosuppressive medication within 14 days before study treatment, except: A. Intranasal, inhaled, topical, or local corticosteroid injections B. Systemic corticosteroids ≤10 mg/day of prednisone or equivalent C. Premedication for hypersensitivity (e.g., CT scan premed) ⑪ Requires mechanical ventilation or vasopressors at enrollment. ⑫ Positive for HIV, active or chronic HBV, active HAV or HCV: A. Known HIV infection B. Positive HBsAg (acute or chronic); HBV DNA PCR required for anti-HBcAb(+) patients.
* EXCEPTION: Isolated anti-HBs with known HBV vaccination
* EXCEPTION: anti-HBc(+), HBsAg(-), anti-HBsAb(-) with negative HBV DNA C. HCV antibody and RNA positive ⑬ Pregnant, breastfeeding, or planning pregnancy during study participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate to Achieve CMV DNA Titer Reduction to < 500 IU/mL | From Week 1 to CMV clearance
  The proportion (%) of patients whose plasma CMV DNA titer decreases to below 500 IU/mL at any point during maribavir treatment, as assessed by local laboratory testing.
Time to Achieve CMV DNA Titer Reduction to < 500 IU/mL | From Week 1 to CMV clearance
  The time (in days) from the initiation of maribavir treatment to the first documented plasma CMV DNA titer of < 500 IU/mL, confirmed by local laboratory testing.
Safety outcomes | From Screening to Week 18
  Adverse events (AEs) will be evaluated in terms of type, frequency, seriousness, and severity, and their relationship to maribavir will be assessed. All AEs will be graded according to the NCI CTCAE criteria, and their causality with study drug will be determined by the investigator.

SECONDARY OUTCOMES:
Rate to Achieve ≥1 log₁₀ Decrease in CMV DNA Titer From Baseline | From Week 1 to CMV clearance
  The proportion (%) of patients who achieve a reduction of ≥1 log₁₀ in plasma CMV DNA titer from baseline (i.e., the time of maribavir initiation), as assessed by local laboratory testing.
Time to Achieve ≥1 log₁₀ Reduction in Plasma CMV DNA Titer From Baseline | From Week 1 to CMV clearance
  The time (in days) from maribavir initiation to the first documented ≥1 log₁₀ decrease in plasma CMV DNA titer from baseline, as assessed by local laboratory testing.
Rate of Breakthrough CMV Disease | From Maribavir Initiation to End of Treatment at 4 Weeks
  The proportion (%) of patients who develop CMV disease during or after maribavir treatment, despite initial virologic control or response.

OTHER OUTCOMES:
Immunity | From Screening Through End of Treatment (Approximately 12 weeks)
  Host immune status will be evaluated using CD4+/CD8+ T-cell counts, serum immunoglobulin levels (IgG, IgA, IgM), and CMV-specific cell-mediated immunity (CMI). CMV-CMI will be assessed at a central lab using the T-SPOT.CMV assay (Oxford Immunotec), which measures interferon-gamma-producing T cells in response to CMV antigens IE-1 and pp65.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No